CLINICAL TRIAL: NCT00664456
Title: A Phase III, Multicenter, Randomized, Controlled Study of Neoadjuvant LHRH-agonist Therapy and Permanent I-125 Implantation With vs. Without Adjuvant LHRH-agonist Therapy in Patients With Untreated Intermediate-risk Prostate Cancer.
Brief Title: Luteinizing Hormone-Releasing Hormone Agonist Therapy and Iodine I 125 Implant in Treating Patients With Previously Untreated Prostate Cancer
Acronym: SHIP0804
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: The Jikei University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRIGU05-01; CDR0000593653 (Other: National Cancer Institute)
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage I prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AHT group (Active Comparator): Randomized patients undergo 3-month neoadjuvant therapy (NHT)within 14 days and receive 9-month adjuvant therapy (AHT) following after Iodine I-125 implantation (TPPB).
  Interventions: Drug: Adjuvant therapy; Drug: Neoadjuvant therapy; Radiation: Brachytherapy（iodine I 125）
- Non-AHT group (Active Comparator): Rondomized patients undergo 3-month neoadjuvant therapy (NHT) within 14 days and receive Iodine I-125 implantation therapy (TPPB). 40 weeks observation is followed under no further treatment.
  Interventions: Drug: Neoadjuvant therapy; Radiation: Brachytherapy（iodine I 125）

INTERVENTIONS:
Drug: Adjuvant therapy — AHT group receives 9 cycle of LHRH-A (goserelin acetate 3.6 mg/4 weeks or leuprorelin acetate 3.75 mg/4 weeks) after Iodine I-125 implantation (TPPB).
  Arms: AHT group
Drug: Neoadjuvant therapy — 3 cycle of LHRH-A (goserelin acetate 3.6mg/4 weeks or leuprorelin acetate 3.75mg/4 weeks).
Radiation: Brachytherapy（iodine I 125） — Undergo Iodine I-125 transperineal prostatic brachytherapy (TPPB).

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Luteinizing hormone-releasing hormone agonists may lessen the amount of androgens made by the body. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving luteinizing hormone-releasing hormone agonist together with an iodine I 125 implant may be an effective treatment for patients with prostate cancer.

PURPOSE: This randomized phase III trial is studying how well giving luteinizing hormone-releasing hormone agonist therapy together with an iodine I 125 implant works with or without additional luteinizing hormone-releasing hormone agonist therapy in treating patients with previously untreated prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the biochemical progression-free survival (PFS), overall survival, clinical PFS, and disease-free survival of patients with previously untreated intermediate-risk prostate cancer treated with neoadjuvant luteinizing hormone-releasing hormone (LHRH) agonist therapy and permanent iodine I 125 implantation with vs without adjuvant LHRH agonist therapy.
* To determine the non-adaptive interval to salvage therapy in patients treated with these regimens.
* To determine the safety of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive neoadjuvant luteinizing hormone-releasing hormone (LHRH) agonist therapy for up to 3 months and undergo permanent iodine I 125 implantation. Patients then receive adjuvant LHRH agonist therapy for up to 9 months.
* Arm II: Patients receive neoadjuvant LHRH agonist therapy and undergo permanent iodine I 125 implantation as in arm I.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed prostate cancer

  * Previously untreated disease
* Intermediate-risk disease, as defined by the following:

  * Clinical stage < T2c
  * Prostate-specific antigen (PSA) ≤ 20 ng/mL
  * Gleason score < 8

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* Leukocyte count ≥ 3,000/uL
* Hemoglobin ≥ 10.0 g/dL
* Platelet count ≥ 100,000/uL
* Serum creatinine ≤ 2.0 mg/dL
* ALT and AST ≤ 100 IU/L
* No other cancer requiring treatment
* No poorly controlled hypertension (i.e., diastolic blood pressure ≥ 120 mm Hg)
* No severe psychiatric disorders, including schizophrenia or dementia
* No poorly controlled diabetes
* Considered appropriate for study participation, as determined by the Principal Investigator or Clinical Investigator

PRIOR CONCURRENT THERAPY:

* No prior drugs for benign prostatic hyperplasia (other than antiandrogen therapy)
* No prior surgery for prostate cancer
* No concurrent steroid drugs (except for ointment)
* No other concurrent antiandrogen therapy

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Biochemical progression-free survival (bPFS) | 7 years
  Interval from the 1st day of treatement to the earliest day on which confirmation of increase in prostate specific antigen (PSA) or death any reason.

SECONDARY OUTCOMES:
Overall survival (OS) | 13.5 years
  Interval from the 1st day of treatment to the earliest day of death any reason.
Clinical progression-free survival | 7 years
  Interval from the 1st day of treatment to the ealiest day on which identification of desease progression or death for any reason.
Disease-specific survival | 7 years
  Interval from the 1st day of treatment to death caused by prostate cancer
Salvage therapy non-adaptive interval | 7 years
  Observational term as salvage therapy non-adaptive interval.
Quality of life (QOL) evaluation | Baseline and Month 60 after TPPB
  QOL assesed by the Japanese version of the SF-8 (the MOS 8 item Short-Form Health Survey), the Japanese version of the Expanded Prostate Cancer Index Composite (EPIC), and the International Prostate Sympton Score (IPSS).
Adverse events (AE) | AE to androgen-deprivation therapy (ADT) within 24 month, AE to 125I-transperineal prostatic brachytherapy (TPPB) within 36 month of the therapy
  The incident propotion of adverse event grade above 3 by National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (NCI-CTCAE v3.0) will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Shin Egawa, MD, PhD, Principal Investigator — The Jikei University School of Medicine
Locations (1):
- The Jikei University School of Medicine, Tokyo, Japan

REFERENCES:
- [Result] Miki K, Kiba T, Sasaki H, Kido M, Aoki M, Takahashi H, Miyakoda K, Dokiya T, Yamanaka H, Fukushima M, Egawa S. Transperineal prostate brachytherapy, using I-125 seed with or without adjuvant androgen deprivation, in patients with intermediate-risk prostate cancer: study protocol for a phase III, multicenter, randomized, controlled trial. BMC Cancer. 2010 Oct 21;10:572. doi: 10.1186/1471-2407-10-572. PMID 20964826
- [Derived] Urabe F, Miki K, Kimura T, Sasaki H, Tashiro K, Iwatani K, Matsukawa A, Aikawa K, Tsusumi Y, Morikawa M, Minato K, Sato S, Takahashi H, Aoki M, Egawa S. Long-term outcomes of radical prostatectomy versus low-dose-rate brachytherapy in patients with intermediate-risk prostate cancer: Propensity score matched comparison. Prostate. 2023 Feb;83(2):135-141. doi: 10.1002/pros.24445. Epub 2022 Sep 29. PMID 36176043
- [Derived] Tabata R, Kimura T, Kuruma H, Sasaki H, Kido M, Miki K, Takahashi H, Aoki M, Egawa S. Do androgen deprivation and the biologically equivalent dose matter in low-dose-rate brachytherapy for intermediate-risk prostate cancer? Cancer Med. 2016 Sep;5(9):2314-22. doi: 10.1002/cam4.820. Epub 2016 Jul 25. PMID 27456710
- [Derived] Sasaki H, Kido M, Miki K, Aoki M, Takahashi H, Dokiya T, Yamanaka H, Fukushima M, Egawa S. Results of central pathology review of prostatic biopsies in a contemporary series from a phase III, multicenter, randomized controlled trial (SHIP0804). Pathol Int. 2015 Apr;65(4):177-82. doi: 10.1111/pin.12260. Epub 2015 Feb 24. PMID 25707702
- [Derived] Sasaki H, Kido M, Miki K, Kuruma H, Takahashi H, Aoki M, Egawa S. Salvage partial brachytherapy for prostate cancer recurrence after primary brachytherapy. Int J Urol. 2014 Jun;21(6):572-7. doi: 10.1111/iju.12373. Epub 2013 Dec 23. PMID 24372730
- [Derived] Kimura T, Kido M, Miki K, Yamamoto T, Sasaki H, Kuruma H, Hayashi N, Takahashi H, Aoki M, Egawa S. Mid-term outcome of permanent prostate iodine-125 brachytherapy in Japanese patients. Int J Urol. 2014 May;21(5):473-8. doi: 10.1111/iju.12347. Epub 2013 Nov 20. PMID 24256329